CLINICAL TRIAL: NCT04106531
Title: Validation of a Novel Patient-Reported Quality of Life Metric "Prolac-10" for Patients Undergoing Medical Therapy for Prolactinoma
Brief Title: Validation of a Quality of Life Metric "Prolac-10"
Acronym: Prolac-10
Status: Terminated | Type: Observational
Why Stopped: Investigator leaving institution
Sponsor: Ohio State University (Other)
Responsible Party: Sponsor
Other Study IDs: 2019H0375
Record Dates: First submitted 2019-09-25; First posted 2019-09-27 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Prolactinoma; Prolactin-Producing Pituitary Tumor; Pituitary Tumor; Prolactinoma Macroadenoma; Prolactinoma Microadenoma
MeSH Terms: conditions — Prolactinoma; Pituitary Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a short-term validation study of a quality of life metric "Prolac-10" for patients diagnosed with a prolactinoma, undergoing new medical therapy.

DETAILED DESCRIPTION:
This is a single-site validation study of a novel quality of life study for patients undergoing medical therapy for prolactinoma. Patients will be consented before starting their medical regimen and complete the "Prolac-10" questionnaire for baseline and will continued to be followed for 13-weeks into their medical care. The primary goal of this study is to validate the novel quality of life questionnaire in terms of sensitivity, repeatability, and consistency. Secondarily, we aim to validate the test-retest characteristics to further validate sensitivity, repeatability, and consistency.

The Prolac-10 metric is Copyright © 2019. The Ohio State University. Modification/derivative rights reserved, all other rights available.

ELIGIBILITY:
Inclusion Criteria:

* Patient has been diagnosed with prolactinoma by use of appropriate blood tests and brain imaging.
* 18 years of age or older
* The subject must in the investigator's opinion, be psychosocially, mentally, and physically able to fully comply with this protocol including the required follow-up visits, the filling out of required forms, and have the ability to understand and give written informed consent

Exclusion Criteria:

* Patient is a prisoner
* Patient is not English speaking
* Patient has been previously treated for prolactinoma
* Patient is pregnant at time of diagnosis and treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study participants will be 18 years or older, diagnosed with a prolactinoma via appropriate laboratory testing and imaging, and will be naive to medical treatment for prolactinoma.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2023-06-13 (Actual); Study Completion 2023-06-13 (Actual)

PRIMARY OUTCOMES:
Validate the "Prolac-10" quality of life metric | 13-weeks post medical therapy start date
  In patients diagnosed with a Prolactinoma, validate the novel quality of life questionnaire, Prolac-10 by testing its sensitivity and internal consistency.

SECONDARY OUTCOMES:
Validate the test-retest characteristics of the Prolac-10 | 13-weeks post medical therapy start date
  Validate the test-retest characteristics of the Prolac-10 to further validate sensitivity, repeatability, and consistency.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Hardesty, MD, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan to share IPD